CLINICAL TRIAL: NCT02019758
Title: Budesonide Versus Fluticasone for Treatment of Eosinophilic Esophagitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-4047; R01DK101856 (NIH)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2019-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide; Fluticasone; trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Viscous Budesonide (OVB) (Active Comparator): Subjects will be treated with OVB at a dose of 1 mg twice daily, and they will also be instructed to use a placebo inhaler identical to the fluticasone MDI, with instructions to swallow 4 puffs twice daily.
  Interventions: Drug: Oral Viscous Budesonide; Drug: Placebo inhaler
- Active Fluticasone MDI (Active Comparator): Subjects will be treated with fluticasone MDI at a dose of 880 mcg twice daily (4 puffs of a 220 mcg inhaler twice daily), and they will also be instructed to take 4 mL twice daily of a placebo slurry of sucralose identical in consistency and taste to the OVB.
  Interventions: Drug: Fluticasone MDI; Drug: Placebo slurry

INTERVENTIONS:
Drug: Oral Viscous Budesonide — Oral Viscous Budesonide - 1 mg/4 mL, 4 mL of slurry twice daily
  Other Names: Pulmicort
  Arms: Oral Viscous Budesonide (OVB)
Drug: Fluticasone MDI — Fluticasone multi-dose inhaler - 4 puffs twice daily (880 mcg, twice daily)
  Other Names: Flovent
  Arms: Active Fluticasone MDI
Drug: Placebo slurry — Slurry of sucralose - 4 mL twice daily
  Other Names: Sucralose
  Arms: Active Fluticasone MDI
Drug: Placebo inhaler — Placebo inhaler - 4 puffs twice daily
  Other Names: Placebo
  Arms: Oral Viscous Budesonide (OVB)

SUMMARY:
Purpose: To determine whether oral viscous budesonide (OVB) or fluticasone metered dose inhaler (MDI) most effectively treats EoE by improving histologic findings and symptoms, which medication provides a more durable treatment response, and whether biomarkers can predict treatment response.

Participants: A total of up to 200 16-80 year old patients with a new diagnosis of eosinophilic esophagitis (EoE) who are referred for upper endoscopy will be consented with a target of 122 randomized.

Procedures: This will be a prospective, randomized, double-blind, double-dummy, clinical trial comparing OVB to fluticasone MDI for treatment of EoE. This overall study design will generate data for all three Aims

DETAILED DESCRIPTION:
This will be a prospective, randomized, double-blind, double-dummy, clinical trial comparing oral viscous budesonide (OVB) to fluticasone metered dose inhaler (MDI) for treatment of EoE. A total of 122 subjects aged 16-80 years old will be randomized in a 1:1 fashion to one of two active treatment arms: OVB + placebo inhaler or fluticasone MDI + placebo slurry.

In the first arm, subjects will be treated with OVB at a dose of 1 mg twice daily, and they will also be instructed to use a placebo inhaler identical to the fluticasone MDI, with instructions to swallow 4 puffs twice daily. The OVB is a slurry equivalent to what is used clinically: 1 mg/4 mL aqueous budesonide mixed with 10 g of sucralose. Rather than asking the subjects to mix the slurry on their own and risk inconsistent formulations, the University of North Carolina (UNC) investigational drug pharmacy (IDP) will provide pre-mixed OVB to all patients. The IDP will also provide placebo inhalers to all patients. The dose for OVB has been chosen because it is the most commonly studied dose, including one prior study led by this Principal Investigator, so we can accurately estimate response rates.

In the second arm, subjects will be treated with fluticasone MDI at a dose of 880 mcg twice daily (4 puffs of a 220 mcg inhaler twice daily), and they will also be instructed to take 4 mL twice daily of a placebo slurry of sucralose identical in consistency and taste to the OVB. The UNC investigational drug pharmacy (IDP) will provide the fluticasone MDIs and pre-mixed placebo slurries to all patients. The dose for fluticasone MDI has been chosen because this is the most commonly used dose in adolescents and adults with EoE, so effect estimates are also available.

For both arms, the slurry will be administered first, the MDI will be administered 15 minutes later, and patients will take nothing by mouth for an additional 30 minutes.

Subjects will receive 8 weeks of treatment and will then be monitored for up to 52 weeks for recurrence of symptoms.

ELIGIBILITY:
Inclusion criteria are as follows:

* Age: 16 - 80 years
* Subject is having a clinically indicated endoscopy for suspicious EoE and has been on twice daily (BID) proton pump inhibitor (PPI) for at least 8 weeks OR New diagnosis of EoE as per consensus guidelines. Cases must have symptoms of dysphagia, persistent esophageal eosinophilia (≥ 15 eosinophils in at least one high-power field) after 8 weeks of treatment with a twice daily proton-pump inhibitor, and other competing causes of esophageal eosinophilia excluded.

Exclusion criteria are as follows:

* Medical instability that precludes safely performing upper endoscopy
* Ongoing or recent symptoms of intestinal bleeding (throwing up blood, passing blood in the stool)
* Concomitant eosinophilic gastroenteritis
* Esophageal narrowing or stricturing that will not allow a standard 9 mm upper endoscopy scope to pass
* Cancer in the esophagus, stomach, or intestine
* Previous esophageal surgery
* Esophageal varices (dilated blood vessels in the esophagus)
* Current use of blood thinners like Plavix or Coumadin that are not stopped prior to endoscopy procedures
* Any corticosteroid exposure within the 4 weeks prior to their baseline endoscopic exam. Exclusionary corticosteroid exposure is defined as any swallowed topical steroids for EoE or systemic steroids for any condition within the four weeks prior to the baseline endoscopy. Corticosteroids used for asthma or intranasal corticosteroids are not an exclusion and are allowable.
* Pregnancy
* Inability to read or understand English

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan S Dellon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Safroneeva E, Cotton CC, Schoepfer AM, Zwahlen M, Woosley JT, Dellon ES. Dilation Modifies Association Between Symptoms and Esophageal Eosinophilia in Adult Patients With Eosinophilic Esophagitis. Am J Gastroenterol. 2020 Dec;115(12):2098-2102. doi: 10.14309/ajg.0000000000000957. PMID 33009060
- [Derived] Dellon ES, Woosley JT, Arrington A, McGee SJ, Covington J, Moist SE, Gebhart JH, Galanko JA, Baron JA, Shaheen NJ. Rapid Recurrence of Eosinophilic Esophagitis Activity After Successful Treatment in the Observation Phase of a Randomized, Double-Blind, Double-Dummy Trial. Clin Gastroenterol Hepatol. 2020 Jun;18(7):1483-1492.e2. doi: 10.1016/j.cgh.2019.08.050. Epub 2019 Sep 6. PMID 31499249
- [Derived] Dellon ES, Woosley JT, Arrington A, McGee SJ, Covington J, Moist SE, Gebhart JH, Tylicki AE, Shoyoye SO, Martin CF, Galanko JA, Baron JA, Shaheen NJ. Efficacy of Budesonide vs Fluticasone for Initial Treatment of Eosinophilic Esophagitis in a Randomized Controlled Trial. Gastroenterology. 2019 Jul;157(1):65-73.e5. doi: 10.1053/j.gastro.2019.03.014. Epub 2019 Mar 11. PMID 30872104

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Viscous Budesonide (OVB): Subjects will be treated with Oral Viscous Budesonide (OVB) at a dose of 1 mg twice daily, and they will also be instructed to use a placebo inhaler identical to the fluticasone MDI, with instructions to swallow 4 puffs twice daily.
  Oral Viscous Budesonide: Oral Viscous Budesonide - 1mg/4 mL, 4 mL of slurry twice daily
  Placebo inhaler: Placebo inhaler - 4 puffs twice daily
- Active Fluticasone Metered Dose Inhaler (MDI): Subjects will be treated with fluticasone Metered Dose Inhaler (MDI) at a dose of 880 mcg twice daily (4 puffs of a 220 mcg inhaler twice daily), and they will also be instructed to take 4 mL twice daily of a placebo slurry of sucralose identical in consistency and taste to the OVB.
  Fluticasone MDI: Fluticasone multi-dose inhaler - 4 puffs twice daily (880 mcg, twice daily)
  Placebo slurry: Slurry of sucralose - 4 mL twice daily
Period: Overall Study
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone Metered Dose Inhaler (MDI)
Started | 65 (64 received intervention; 1 did not receive intervention) | 64 (63 received intervention; 1 did not receive intervention)
Received Intervention | 64 | 63
Did Not Receive Intervention | 1 | 1
Lost to Follow-up | 8 (8 were lost to follow-up and did not undergo week 8 endoscopy or other outcome assessments) | 8 (8 were lost to follow-up and did not undergo week 8 endoscopy or other outcome assessments)
Completed | 56 | 55 (8 were lost to follow-up and did not undergo week 8 endoscopy or other outcome assessments)
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Oral Viscous Budesonide (OVB): Subjects will be treated with OVB at a dose of 1 mg twice daily, and they will also be instructed to use a placebo inhaler identical to the fluticasone MDI, with instructions to swallow 4 puffs twice daily.
  Oral Viscous Budesonide: Oral Viscous Budesonide - 1mg/4 mL, 4 mL of slurry twice daily
  Placebo inhaler: Placebo inhaler - 4 puffs twice daily
- Total: Total of all reporting groups
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (19.1) | 39.0 (14.5) | 38.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 40 | 44 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 63 | 63 | 126
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 64 | 129

OUTCOME MEASURES:

1. Primary Outcome: Post-Treatment Maximum Eosinophil Count (Aim 1)
Description: To determine whether viscous budesonide is more effective than fluticasone MDI for improving post-treatment maximum esophageal eosinophil counts (measured in eosinophils per high powered field (eos/hpf)) in patients with eosinophilic esophagitis (EoE). The mean post-treatment maximum eosinophil count will be compared between the OVB and MDI groups using a two-sample t-test.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: eosinophils per high-power field
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 56 | 55
eosinophils per high-power field | 14.7 (29.0) | 20.9 (34.3)
Statistical Analysis 1: Comparison: Oral Viscous Budesonide (OVB) vs Active Fluticasone MDI; The mean post-treatment maximum eosinophil count will be compared between the OVB and MDI groups using a two-sample t-test; Test type: Superiority; p = 0.31, t-test, 2 sided

2. Primary Outcome: Post-treatment Dysphagia Score (Aim 1)
Description: To determine whether viscous budesonide is more effective than fluticasone MDI for improving dysphagia (measured by the Daily Symptoms Questionnaire (DSQ)) in patients with EoE. The mean DSQ scores will be compared between the OVB and MDI groups using a two-sample t-test. The DSQ is a dysphagia severity score which ranges from 0-84, with higher numbers indicating more severe symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 56 | 55
score on a scale | 4.8 (7.3) | 4.2 (7.5)
Statistical Analysis 1: Comparison: Oral Viscous Budesonide (OVB) vs Active Fluticasone MDI; The mean DSQ scores will be compared between the OVB and MDI groups using a two-sample t-test; Test type: Superiority; p = 0.70, t-test, 2 sided

3. Secondary Outcome: Post-treatment Endoscopic Severity (Aim 1)
Description: Endoscopic severity will be quantified using the EoE Endoscopic Reference Score (EREFS) and compared between the two treatment arms. EREFS is a validated endoscopic severity score of key EoE endoscopic features (exudates, rings, edema, furrows, and strictures), and ranges from 0-9 with higher scores indicating higher endoscopic severity.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 56 | 55
score on a scale | 2.1 (1.7) | 2.8 (2.2)

4. Secondary Outcome: Percentage of Participants With Histologic Response of <15 Eos/Hpf
Description: Percentage with histologic response, with response defined as <15 eos/hpf, will be compared between groups
Time Frame: 8 weeks
Measure: Number; unit: Percent responders
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 56 | 55
Percent responders | 71 | 64

5. Secondary Outcome: Post-treatment Symptom Severity (Aim 1)
Description: Post-treatment symptoms severity will be assessed with the EoE Symptom Activity Index (EEsAI), a validated dysphagia severity measure. The EEsAI ranges from 0-100, with higher scores indicating more severe symptoms; symptom remission is defined by a score <20.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 56 | 55
score on a scale | 22.1 (18.9) | 28.0 (20.4)

6. Secondary Outcome: Post-treatment Medication Compliance (Aim 1)
Description: Medication compliance as measured by the percentage of medication appropriately used in each arm. For the slurry, this percentage is calculated after measuring the residual volume. For the inhaler, this percentage is calculated after measured using the residual weight.
Time Frame: 8 weeks
Measure: Number; unit: Percentage of medication used
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 56 | 55
Percentage of medication used | 87 | 85

7. Secondary Outcome: Median Number of Days Until Symptom Recurrence (Aim 2)
Description: To test whether OVB results in less symptomatic recurrence than fluticasone MDI, the median number of days until symptom occurrence will be quantified between treatment end (week 8) and recurrent symptoms or study end (week 60) as the time of interest. Hazard ratio will be calculated using Cox proportional modeling.
Time Frame: Symptom recurrence or 1 year after completing the initial 8 week treatment
Population: This population reflects only those patients who achieved histologic remission (<15 eosinophils per high-power field) after the blinded phase, entered the observation phase, and had symptom outcome data.
Measure: Median (Standard Error); unit: Days
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 33 | 25
Days | 263 (42.0) | 224 (66.3)
Statistical Analysis 1: Comparison: Oral Viscous Budesonide (OVB) vs Active Fluticasone MDI; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.52 to 2.08]

8. Secondary Outcome: Number of Subjects With Histologic Recurrence, Defined as ≥15 Eosinophils Per High-power Field, at Follow-up Endoscopy.
Description: To test whether OVB results in less histologic recurrence than fluticasone MDI, the number of subjects with ≥15 eosinophils per high-power field at follow-up endoscopy in each group will be compared using chi-square.
Time Frame: Symptom recurrence or 1 year after completing the initial 8 week treatment
Population: This population reflects only those patients who achieved histologic remission (<15 eosinophils per high-power field) after the blinded phase, entered the observation phase, and had endoscopic and histologic data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 25 | 25
Participants | 22 | 17
Statistical Analysis 1: Comparison: Oral Viscous Budesonide (OVB) vs Active Fluticasone MDI; Test type: Superiority; p < 0.001, Chi-squared

9. Secondary Outcome: Mean Endoscopic Severity Score at Recurrence (Aim 2)
Description: Measurement of endoscopic severity, using the EoE Endoscopic Reference Score (EREFS) measure, at the time of recurrence. EREFS is a validated endoscopic severity score of key EoE endoscopic features (exudates, rings, edema, furrows, and strictures), and ranges from 0-9 with higher scores indicating higher endoscopic severity.
Time Frame: Symptom recurrence or 1 year after completing the initial 8 week treatment
Population: This population reflects only those patients who achieved histologic remission (<15 eosinophils per high-power field) after the blinded phase, entered the observation phase, and had endoscopic and histologic outcome data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 25 | 25
score on a scale | 4.8 (1.7) | 4.3 (2.0)
Statistical Analysis 1: Comparison: Oral Viscous Budesonide (OVB) vs Active Fluticasone MDI; Test type: Superiority; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Mean Peak Eosinophil Count (Aim 2)
Description: This will assess the mean peak level of esophageal eosinophilia on biopsy (measured in peak eosinophil count - eos/hpf) at the time of recurrence
Time Frame: Symptom recurrence or 1 year after completing the initial 8 week treatment
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: eosinophils per high-power field
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
Number analyzed (Participants) | 25 | 25
eosinophils per high-power field | 71.8 (52.9) | 35.0 (29.4)
Statistical Analysis 1: Comparison: Oral Viscous Budesonide (OVB) vs Active Fluticasone MDI; Test type: Superiority; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 weeks over the initial treatment period.
Arm/Group | Oral Viscous Budesonide (OVB) | Active Fluticasone MDI
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/65 | 1/64
Other Adverse Events (participants affected / at risk) | 10/65 | 15/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Viscous Budesonide (OVB) (N=65) | Active Fluticasone MDI (N=64)
Food impaction (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Viscous Budesonide (OVB) (N=65) | Active Fluticasone MDI (N=64)
esophageal candidiasis (Gastrointestinal disorders) | 8 | 10
oral candidiasis (Gastrointestinal disorders) | 2 | 1
sore throat (Gastrointestinal disorders) | 0 | 2
chest pain (Cardiac disorders) | 0 | 1
pneumonia (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02019758/Prot_SAP_000.pdf